CLINICAL TRIAL: NCT05482529
Title: A Prospective Study of Integrative Omics Analysis for Colorectal Cancer and Metastasis
Brief Title: Integrative Omics Analysis for Colorectal Cancer and Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: fan li (Other)
Responsible Party: Sponsor-Investigator, fan li, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: IOACCM
Record Dates: First submitted 2022-05-04; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer
Keywords: Integrative omics; colorectal cancer; distant metastasis; prognostic analysis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Colorectal cancer (CRC), adjacent colon, lymph nodes (LN) along colons, metastasis (DM), and adjacent of metastasis ,lymph nodes (LM) along metastasis ,and peripheral blood mononuclear cells (PBMC)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer with metastasis: colorectal cancer patients with at least one distant metastasis(liver, lung)
  Interventions: Other: Integrative omics

INTERVENTIONS:
Other: Integrative omics — Integrative omics such as RNA-sequencing,ATAC-seq(Assay for Transposase-Accessible Chromatin using sequencing), CUT&Tag（ Cleavage Under Targets and Tagmentation）to analyze and predict candidate biomarkers of colorectal cancer and distant metastasis.

SUMMARY:
The pathogenesis of Colorectal cancer (CRC) metastasis remains unclear.We collect clinical data from our center and use Integrative omics to analyze and predict candidate biomarkers of colorectal cancer and distant metastasis.

DETAILED DESCRIPTION:
Colorectal cancer (CRC), one of the most common malignant cancer around the world, CRC patients with distant metastasis. However, the pathogenesis of metastasis remains unclear. Integrative omics have begun to enable personalized medicine at an extraordinarily detailed molecular level. All patients with colorectal cancer and metastasis in our center who meet the inclusion criteria and exclusion criteria will be enrolled. The specimen collected by surgery and clinical data will be collected . We use Integrative omics such as RNA-sequencing,ATAC-seq(Assay for Transposase-Accessible Chromatin using sequencing), CUT&Tag（ Cleavage Under Targets and Tagmentation）to analyze and predict candidate biomarkers of colorectal cancer and distant metastasis. This study will contribute to understanding the molecular mechanism of CRC metastasis in depth and contribute to the discovery of new appropriate molecular diagnostic and therapeutic targets, and more accurately prognose long term outcome in patients with CRC.

ELIGIBILITY:
Inclusion Criteria:

* colorectal adenocarcinoma by biopsy。
* at least 1 metastasis lesion comfirmed by at least 1 kind of imaging examination (CT, MRI and PET-CT )

Exclusion Criteria:

* recent diagnosis with other malignancies
* can not tolerate the surgery
* history of serious mental illness
* pregnancy or lactating women
* the researchers believe the patients should not enrolled in

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with colorectal cancer and metastasis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | 3 years after surgery
  the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
disease free survival rate | 3 years after surgery
  the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.

SECONDARY OUTCOMES:
Quality of life outcomes evaluation(QLQ-CR38) | 0- 2 years after surgery
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (HRQoL).The General quality of life quality of life Questionnaires of Colorectal Cancer-38(QLQ-CR38) are used to evaluate the Quality of life outcomes. Items are scored on a four-point scale from 1("not at all) to 4 ("very much"). Raw scores are aggregated and converted to a linear scale ranging from 0 to 100, with higher scores representing a higher level of functioning or a higher level of symptoms
Quality of life outcomes evaluation(QLQ-C30) | 0- 2 years after surgery
  We examine before operation, 3 months after, 6 months after, 12 months after, 24 months after operation, by questionnaires (HRQoL).The General quality of life Quality of life Questionnaires of Cancer-30 (QLQ-C30) are used to evaluate the Quality of life outcomes. Items are scored on a four-point scale from 1("not at all) to 4 ("very much"). Raw scores are aggregated and converted to a linear scale ranging from 0 to 100, with higher scores representing a higher level of functioning or a higher level of symptoms
R0 resection rate | 2 weeks after surgery
  The R0 resection rate by pathology outcome of specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Daping hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided